CLINICAL TRIAL: NCT06255210
Title: Efficacy and Safety of Induction Chemotherapy for Olfactory Neuroblastoma: a Prospective Umbrella Clinical Study
Brief Title: Efficacy and Safety of Induction Chemotherapy for Olfactory Neuroblastoma (ESICON)
Acronym: ESICON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hongmeng Yu (Other)
Responsible Party: Sponsor-Investigator, Hongmeng Yu, Professor, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONB-NACT-V1
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Olfactory Neuroblastoma
Keywords: Induction Chemotherapy
MeSH Terms: conditions — Esthesioneuroblastoma, Olfactory

STUDY DESIGN:
Intervention Model Description: umbrella design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction chemotherapy in different subtypes of olfactory neuroblastoma (Experimental): Induction chemotherapy based on pathological molecular subtypes of olfactory neuroblastoma.
  ① According to the immunohistochemical results of the pathological report, patients with Ki-67 index ≥ 25% were treated with two weeks of gemcitabine+platinum based chemotherapy regimen;
  ② According to the immunohistochemical results of the pathological report, patients with Ki-67 index <25% were treated with a basic chemotherapy regimen of cyclophosphamide+etoposide+cisplatin (CEP regimen);
  According to the progression of the patient's disease, the combination of other chemotherapy/small molecule drugs/targeted drugs can be considered;
  Interventions: Drug: Gemcitabine+Cisplatin(GP); Cyclophosphamide+Etoposide+Cisplatin(CEP)

INTERVENTIONS:
Drug: Gemcitabine+Cisplatin(GP); Cyclophosphamide+Etoposide+Cisplatin(CEP) — When the Ki67% index of the tumor is ≥ 25%, patients were treated with the GP regimen for induction chemotherapy; When the Ki67% index of the tumor is < 25%, patients were treated with the CEP regimen for induction chemotherapy.

SUMMARY:
The goal of this clinical trial is to learn about the induction chemotherapy efficacy in olfactory neuroblastoma. The main question it aims to answer is: wether olfactory neuroblastoma patients with different pathology subtypes apply to different induction chemotherapy schemes. Participants will be treated with different chemotherapy schemes, to evaluate the tumor remission rate and long term survival.

DETAILED DESCRIPTION:
This study included patients with olfactory neuroblastoma who were pathologically diagnosed and met the criteria. According to molecular profiles, two different induction chemotherapy schemes were used to evaluate the tumor remission rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed olfactory neuroblastoma;
2. Age ≥ 18 years old;
3. Dulguerov stage T2-T4;
4. Patients who signed the informed consent forms;
5. No distant metastasis.

Exclusion Criteria:

1. Patients with uncontrolled concurrent diseases that the researchers believe will interfere with treatment;
2. Any situation in which the patient may interfere with the compliance or safety during the study;
3. Severe neurological or mental illness, including dementia and seizures;
4. Uncontrolled active infection;
5. Pregnant or lactating women;
6. Persons without personal freedom and independent capacity for civil conduct;
7. Other situations that are not suitable for joining the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate(ORR) | 3 to 12 weeks after completion of induction chemotherapy
  According to RECIST1.1 criteria, complete remission (CR) and partial remission (PR)

SECONDARY OUTCOMES:
Pathological complete remission(pCR) rate after induction chemotherapy. | about 4 weeks after surgical resection, up to 12 weeks
  pCR rate refers to the probability that no tumor cells was found during pathological diagnosis of tumor sample of surgical treatment after induction chemotherapy, in all patients who have been enrolled in the group.
The rate of surgical pathology negative margin | about 4 weeks after surgical resection, up to 12 weeks
  During the surgery after induction chemotherapy, 4-6 surgical margins were retrieved for each patient. The rate of surgical pathology negative margin refers to the probability that pathological examination showed no tumor cells in all surgical margins, among all patients who have been enrolled in the group.
2-year overall survival (OS) rate | 2 years (24 months)
  The 2-year OS rate refers to the proportion of alive patients 2 years after enrollment, analyzed using the Kaplan Meier method.
Rate of treatment related side effects | 2 years (24 months)
  Refers to the incident rate of side effects related to the prescribed treatment during the induction chemotherapy and the whole follow-up duration. Treatment-related side effects were evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Hongmeng Yu, Prof., Principal Investigator — Eye & ENT Hospital, Fudan University; Xicai Sun, MD, Study Director — Eye & ENT Hospital, Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Study Protocol, Informed Consent Form (ICF), Clinical Study Report (CSR) and Analytic Code were to be shared on request.

REFERENCES:
- [Background] Svane-Knudsen V, Jorgensen KE, Hansen O, Lindgren A, Marker P. Cancer of the nasal cavity and paranasal sinuses: a series of 115 patients. Rhinology. 1998 Mar;36(1):12-4. PMID 9569435
- [Background] Limaiem F, Das JM. Esthesioneuroblastoma. 2023 Jun 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK539694/ PMID 30969516
- [Background] Kim N, Lee CG, Kim EH, Kim CH, Keum KC, Lee KS, Chang JH, Suh CO. Patterns of failures after surgical resection in olfactory neuroblastoma. J Neurooncol. 2019 Jan;141(2):459-466. doi: 10.1007/s11060-018-03056-0. Epub 2018 Nov 30. PMID 30506150
- [Background] Dulguerov P, Allal AS, Calcaterra TC. Esthesioneuroblastoma: a meta-analysis and review. Lancet Oncol. 2001 Nov;2(11):683-90. doi: 10.1016/S1470-2045(01)00558-7. PMID 11902539
- [Background] Classe M, Yao H, Mouawad R, Creighton CJ, Burgess A, Allanic F, Wassef M, Leroy X, Verillaud B, Mortuaire G, Bielle F, Le Tourneau C, Kurtz JE, Khayat D, Su X, Malouf GG. Integrated Multi-omic Analysis of Esthesioneuroblastomas Identifies Two Subgroups Linked to Cell Ontogeny. Cell Rep. 2018 Oct 16;25(3):811-821.e5. doi: 10.1016/j.celrep.2018.09.047. PMID 30332658